CLINICAL TRIAL: NCT06183879
Title: Comparison of Expandable and Fixed Size Cryoballoon for the Treatment of Paroxysmal Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vedran Velagic, MD, PhD, Assistant Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolarvsAFA
Record Dates: First submitted 2023-11-20; First posted 2023-12-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to two different cryoballoon devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medtronic 4th gen balloon (Active Comparator): Cryoballoon pulmonary vein isolation with Medtronic Artic Front Advance Pro 28 mm fixed size cryoballoon
  Interventions: Device: cryoballoon pulmonary vein isolation (Medtronic 4th gen balloon)
- Boston 2nd gen balloon (Active Comparator): Cryoballoon pulmonary vein isolation with Polar X Fit, 28 to 31 mm expandable cryoballoon
  Interventions: Device: cryoballoon pulmonary vein isolation (Boston 2nd gen balloon)

INTERVENTIONS:
Device: cryoballoon pulmonary vein isolation (Medtronic 4th gen balloon) — Standard of care cryoballoon pulmonary vein isolation with Medtronic 4th gen balloon
  Arms: Medtronic 4th gen balloon
Device: cryoballoon pulmonary vein isolation (Boston 2nd gen balloon) — Standard of care cryoballoon pulmonary vein isolation with Boston 2nd gen balloon
  Arms: Boston 2nd gen balloon

SUMMARY:
The goal of this clinical trial is to compare two different, market approved, cryoballoon devices for the treatment of paroxysmal atrial fibrillation (AF).

The main aims of the study are:

* to compare the efficacy of two ablation devices (acute and 1 year success rates)
* to compare the procedural characteristics (procedure duration, fluoroscopy duration, ablation time
* to compare the complication rates

Participants who have indication for cryoballoon ablation of AF will be randomized in 1:1 fashion to older fixed size cryoballoon and newer expandable cryoballoon. Standard of care cryoballoon procedure will be performed alongside with standard postprocedural follow-up.

• to compare the complication rates

Participants who have indication for cryoballoon ablation of AF will be randomized in 1:1 fashion to older fixed size cryoballoon and newer expandable cryoballoon.

DETAILED DESCRIPTION:
Patients suffering from paroxysmal atrial fibrillation who are scheduled (independently of this study) for cryoballoon pulmonary vein isolation will be informed about the study and potential risks. All patients who give written informed consent will be randomized to 4th generation Artic Front Advance Pro device (fixed size balloon of 28 mm) and Polar X Fit device (28-31 mm expandable balloon). The ablation procedure will be performed in standard of care fashion. Also, standard postprocedural follow up of the patients will be scheduled with outpatient clinic visits and 24-hour Holters and 3, 6 and 12 months, and yearly thereafter. Extra visits will be scheduled in the case of symptoms/palpitations.

Standard patient and procedural data will be collected alongside with the information obtained in the follow up.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation
* patient scheduled for cryoballoon pulmonary vein isolation regardless of this study

Exclusion Criteria:

* unwilling to sing the informed consent Left atrium size > 55 mm Uncontrolled heart failure (NYHA III-IV) Intracardiac thrombi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
acute success | 1 week
  successful pulmonary vein isolation, as percentage of all pulmonary veins treated
mid term success | 1 year. Outpatient visits planned on 90, 180 and 360 days.
  number of patients free from atrial arrhythmia (atrial fibrillation detected by ECG or Holter monitors on follow up visits)

SECONDARY OUTCOMES:
procedure duration | 1 week
  duration of the procedure in minutes
fluoroscopy time | 1 week
  fluoroscopy time (minutes)
complications | 1 year
  number of minor (groin hematoma, chest pain, etc) or major complications (tamponade, phrenic nerve palsy, etc)
ablation time | 1 week
  cumulative time of cryo applications in seconds
radiation dosage | 1 week
  radiation dosage (microGrays-m2)

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - KB Dubrava, Zagreb, Please Select
  - KBC Zagreb, Zagreb

IPD SHARING:
Plan to Share IPD: No